CLINICAL TRIAL: NCT00495209
Title: Pre-Surgical Qigong Therapy for Women With Breast Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2005-0876
Record Dates: First submitted 2007-06-28; First posted 2007-07-02 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: Complementary and Alternative Medicine; Breast Cancer; Qigong; Medical Qigong; External Qi Therapy; EQT
MeSH Terms: conditions — Breast Neoplasms | interventions — Qigong

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Qigong: Pre-surgical Qigong therapy for women with breast cancer
  External Qi Therapy = EQT
  Interventions: Other: Qigong

INTERVENTIONS:
Other: Qigong — EQT daily for 5 consecutive days prior to surgery.
  Other Names: Bioenergy Therapy; External Qi Therapy; EQT

SUMMARY:
The use of complementary and alternative medicine (CAM) in the United States has increased dramatically in the past 10 years. Nowhere is this trend more apparent than when one examines CAM use by patients diagnosed with cancer. As with the general population, patients with cancer typically use CAM-based modalities alongside their conventional cancer treatments. Patients are often seeking a holistic approach to managing and preventing disease. Although most patients will combine alternative approaches with conventional medicine, some patients do in fact decline curative conventional treatments in favor of more non-toxic alternative approaches. One such approach that patients combine with conventional medicine or use in place of conventional medicine is qigong.

Qigong is a bioenergy therapy with a long history of therapeutic use for many diseases, including cancer. Preliminary experiments and a review of the literature show that qigong might improve the outcome for cancer patients. However, none of this research has been confirmed in the peer-reviewed Western scientific literature. Although it is unlikely that EQT will result in significant decreases in tumor size, patients are using qigong either as a complementary approach, and sometimes even in place of conventional medicine, it is, therefore, important for us to determine whether there is any merit to this treatment modality. The goal of this pilot trial is to examine one form of medical qigong (external qi therapy (EQT)) to determine feasibility. In an exploratory nature we will also examine any changes in tumor size in women with breast cancer who are awaiting surgery.

DETAILED DESCRIPTION:
Some research has been done on the human body to learn about how it may exist within an electromagnetic (energy with electric and magnetic parts) field. Some research has shown that changing the form of this field may have an effect on cell growth.

You will be asked to complete 3 questionnaires that ask about your quality of life (QOL), your physical functioning, and any symptoms you may be having. The questionnaires will take about 15 to 20 minutes to complete. You will also have a physical exam. If you have had mammogram and ultrasound less than one week after your core biopsy, you will need to have a repeat mammogram and ultrasound to check the size of your tumor.

You will then be scheduled for a total of 5 EQT sessions (1 session per day for 5 consecutive days). You will meet with an expert in EQT (qigong master) to conduct the sessions. During each session, the qigong master will send forth qi (energy) focused toward helping to improve patients' physical and mental functioning. The qigong master will do this by placing his hands over the affected area and emitting his energy into your body. He will not touch you, but will say a few words. These comments will be spoken in Chinese and may be translated into English by a translator. The sessions may be conducted in a group setting. After each session, you will have a physical exam. Each session will last about 30 minutes.

Once you have completed all the sessions, you will have a follow-up visit. During this visit, you will have a physical exam and a mammogram and ultrasound to check the size of your tumor. You will also be asked to complete 3 more questionnaires that will ask the same questions as before. The questionnaires will take about 15 to 20 minutes to complete.

In order to find out if women are willing to have EQT, researchers will keep track of how many people are asked to join the study and how many decide to participate. If you consent to participate, the study staff will keep track of the EQT sessions you attend, if you complete the questionnaires, and if you provide the optional blood samples.

Your participation in this study will be over after your follow-up visit.

This is an investigational study. The baseline mammogram and ultrasound are standard of care. All questionnaires and the follow-up mammogram and ultrasound are for research purposes. Up to 10 patients will take part in this study. All will be enrolled at M. D. Anderson or Fudan University Cancer Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed and intact invasive ductal carcinoma
2. Women with a single measurable mass less than or equal to 3 cm
3. Women who are awaiting the surgical removal of breast cancer
4. Surgery is scheduled at least 2 weeks from the time of recruitment
5. Willing to come to MDACC or Fudan University Cancer Hospital (FUCH) for 5 consecutive days to receive the EQT
6. 18 years of age or older because the assessment tools are not validated for use in minors.

Exclusion Criteria:

1. Women with lobular carcinoma
2. Prior or planned neoadjuvant treatment with chemotherapy or radiotherapy
3. Evidence of metastatic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with breast cancer who are awaiting surgery.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2006-07-26 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of conducting external qigong in women with breast cancer awaiting surgery | 3 Years

SECONDARY OUTCOMES:
Initial efficacy of external qi therapy (EQT) as measured by tumor size | Baseline to end of treatment (5 days)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org